## Testing a Self-affirmation Intervention for Use in a Mobile Application ${\tt January~1,~2018}$

## **Smoking Attitudes**

Welcome to "Smoking attitudes," a web-based research study that explores people's attitudes and beliefs about smoking. Before taking part in this study, please read the consent form below and click on the "I Agree" button at the bottom of the page if you understand the statements and freely consent to participate in the study.

## **Consent Form**

You are being invited to take part in a research study. It is up to you to decide whether to take part in this study. Please take time to read the following information carefully. The purpose of this study is to explore individuals' attitudes and beliefs about cigarette smoking. You may be asked to answer some questions about your opinions or about your past behavior. You will read a short message and provide your reaction to this information. The study is being conducted by Dr. Jennifer Taber of Kent State University and Drs. Erika Waters and Amy McQueen of Washington University in St. Louis. This study has been approved by the Kent State University Institutional Review Board. No deception is involved, and the study involves no more than minimal risk to participants (i.e., the level of risk encountered in daily life). You may skip any questions you prefer not to answer.

Participation in this study should take no longer than 20 minutes and is strictly anonymous. In this study, you will be asked to read a short message about smoking and then complete questions about your own attitudes and beliefs about smoking. After you answer these questions, you will be asked to answer a few questions about yourself. You will receive your standard incentive for completing the study.

Potential Risks: The procedures described above are thought to involve minimal risks to research participants. You may become concerned about your risk of developing a smoking-related disease after reading and answering questions about this topic. At the end of the study, you will be given information about some resources that you may use if you have further questions about your cigarette smoking or are interested in changing your behavior.

Benefits and Compensation: No direct physical, health, psychological or social benefits to participants are expected to result from participation in this study. However, your responses will provide valuable information about the beliefs people have about smoking that may be useful to researchers and practitioners interested in how to help people quit smoking. You will receive the standard reward points you usually receive from Survey Sampling International for a survey that is no more than 20 minutes in duration.

Confidentiality: All responses are treated as confidential, and in no case will responses from individual participants be identified. Rather, all data will be pooled and published in aggregate form only. This study is anonymous as are your responses. Only the researcher and members of her study team will have access to this information.

Withdrawal and termination from the study: Participation is voluntary, refusal to take part in the study involves no penalty or loss of benefits to which participants are otherwise entitled, and

participants may withdraw from the study at any time without penalty or loss of benefits to which they are otherwise entitled. You may skip any questions you prefer not to answer.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>. This website will not include information that can identify you. At most, the website will include a summary of results. This is a public website that you can visit and search at any time.

If participants have further questions about this study or their rights, or if they wish to lodge a complaint or concern, they may contact the principal investigator, Jennifer Taber, PhD., by email (<a href="mailto:itaber1@kent.edu">itaber1@kent.edu</a>) or phone (330-672-3783) or the Kent State University Institutional Review Board (330-672-2704).

If you are 21 years of age or older, understand the statements above, and freely consent to participate in the study, click on the "I Agree" button to begin the study.

